CLINICAL TRIAL: NCT01715246
Title: Clinical Safety of a New Infant Starter Formula Containing 2 Human Milk Oligosaccharides (HMOs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11.26.INF
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: healthy babbies; infant formula; growth; HMO
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Starter infant formula without HMO (Placebo Comparator): Volumes of feed depend on age, weight and appetite.
  Interventions: Other: Infant Formula
- Starter infant formula with 2 HMOs (Active Comparator): Volumes of feeds depend on age, weight and appetite
  Interventions: Other: Infant Formula
- Breasfed reference group (No Intervention)

INTERVENTIONS:
Other: Infant Formula
  Arms: Starter infant formula with 2 HMOs; Starter infant formula without HMO

SUMMARY:
The primary objective of this clinical study is to show that infants fed a standard starter infant formula with 2 Human Milk Oligosaccharides (HMOs) have a growth in line with infants fed a standard starter infant formula without HMOs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy babies
* Full term babies (37 weeks ≤ gestation ≤ 42 weeks)
* birth weight between 2500 g- 4500g
* Having obtained the baby's legal representative's informed consent.
* FF groups:

babies aged between birth and 14 days, exclusively formula-fed at time of enrollment, whose mother independently elected, before enrollment, not to breastfeed

• BF group: babies aged 3 months (+/- 5 days), exclusively breastfed since birth.

Exclusion Criteria:

* Congenital illness or malformation that may affect growth
* Significant pre-natal and/or serious post-natal disease before enrollment (by medical decision)
* Minor parent(s)
* Newborn whose parents / caregivers cannot be expected to comply with study procedures
* Currently participating or having participated in another clinical trial since birth, except for BF group, where vaccines studies are allowed.

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 176 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Growth | 4 months of life
  child growth (body weight) from enrollment to 4 months of age

SECONDARY OUTCOMES:
Growth | 6 and 12 months of age
Digestive tolerance (stool charecteristics, bowel movements,behavior patterns) | every month during 6 months
  Parents are asked to complete a diary on digistive tolerance of their child
Product compliance (quantity of formula in ml consumed on the 3 days before visit) | every month for 6 months
  Parents are asked to complete a diary on the product compliance
Morbidity | ongoing for 1 year
Stool microbiota | 3 and 12 months of age
Gene expression | 3 and 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni CORSELLO, Principal Investigator — Dipartimento Materno Infantile, Palermo; Philippe ALLIET, Principal Investigator — Kinderartsenpraktijk, Hasselt, Belgium
Locations (2):
- Kinderartsenpraktijk, Hasselt, Belgium
- Dipartimento Materno Infantile, Palermo, Italy

REFERENCES:
- [Derived] Tarrant I, Finlay BB. Human milk oligosaccharides: potential therapeutic aids for allergic diseases. Trends Immunol. 2023 Aug;44(8):644-661. doi: 10.1016/j.it.2023.06.003. Epub 2023 Jul 11. PMID 37438187
- [Derived] Dogra SK, Martin FP, Donnicola D, Julita M, Berger B, Sprenger N. Human Milk Oligosaccharide-Stimulated Bifidobacterium Species Contribute to Prevent Later Respiratory Tract Infections. Microorganisms. 2021 Sep 12;9(9):1939. doi: 10.3390/microorganisms9091939. PMID 34576834
- [Derived] Berger B, Porta N, Foata F, Grathwohl D, Delley M, Moine D, Charpagne A, Siegwald L, Descombes P, Alliet P, Puccio G, Steenhout P, Mercenier A, Sprenger N. Linking Human Milk Oligosaccharides, Infant Fecal Community Types, and Later Risk To Require Antibiotics. mBio. 2020 Mar 17;11(2):e03196-19. doi: 10.1128/mBio.03196-19. PMID 32184252
- [Derived] Puccio G, Alliet P, Cajozzo C, Janssens E, Corsello G, Sprenger N, Wernimont S, Egli D, Gosoniu L, Steenhout P. Effects of Infant Formula With Human Milk Oligosaccharides on Growth and Morbidity: A Randomized Multicenter Trial. J Pediatr Gastroenterol Nutr. 2017 Apr;64(4):624-631. doi: 10.1097/MPG.0000000000001520. PMID 28107288